CLINICAL TRIAL: NCT01961427
Title: Dose and Response of Dietary and Inorganic Nitrate in Healthy and Active Men
Brief Title: Dose and Response of Dietary Nitrate in Healthy and Active Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-12
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: dietary nitrate; beetroot juice; exercise performance; oxygen consumption
MeSH Terms: interventions — sodium nitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- sodium Nitrate 12mmol (Active Comparator): Ingestion of a solution of inorganic nitrate, dosage: 12mmol
  Interventions: Dietary Supplement: sodium nitrate
- sodium Nitrate (6mmol) (Active Comparator): ingestion of inorganic nitrate (6mmol solution)
  Interventions: Dietary Supplement: sodium nitrate
- sodium nitrate 3mmol (Active Comparator): ingestion of inorganic nitrate (3mmol solution)
  Interventions: Dietary Supplement: sodium nitrate
- sodium nitrate (0mmol) (Active Comparator): Ingestion of water as a placebo
  Interventions: Dietary Supplement: sodium nitrate
- Beetroot juice (12mmol) (Active Comparator): ingestion of 170ml of concentrated beetroot juice (12mmol)
  Interventions: Dietary Supplement: Beetroot juice
- beetroot juice (6mmol) (Active Comparator): ingestion of 85ml concentrated beetroot juice (6mmol)
  Interventions: Dietary Supplement: Beetroot juice
- Beetroot juice (3mmol) (Active Comparator): Ingestion of 42.5ml of concentrated beetroot juice (3mmol)
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: sodium nitrate — Ingestion of 3mmol, 6mmol and 12mmol sodium nitrate
  Other Names: Inorganic nitrate
  Arms: sodium Nitrate (6mmol); sodium Nitrate 12mmol; sodium nitrate (0mmol); sodium nitrate 3mmol
Dietary Supplement: Beetroot juice — concentrated beetroot juice (dosage 3mmol, 6mmol and 12mmol)
  Other Names: Biotta beetroot juice shot
  Arms: Beetroot juice (12mmol); Beetroot juice (3mmol); beetroot juice (6mmol)

SUMMARY:
It was shown by some researchers that dietary nitrate such as beet root juice can lower oxygen consumption in men and act as a performance enhancing supplement.

It was not shown, what the optimal dosage is and if there is any difference in oxygen consumption comparing beet root juice and inorganic nitrate.

Therefore, the aim of the study is to conduct a study ingesting different sodium nitrate and beet root juice dosages. We would measure nitrate and nitrite concentrations in the blood at different time points and the subjects have to perform an exercise test measuring oxygen consumption 3 hours after the ingestion of nitrate.

DETAILED DESCRIPTION:
1. The subjects have to ingest 7 different dosages of either beetroot juice or sodium nitrate on seven different occasions. Every hour a blood withdrawal is taken to measure nitrate and nitrite concentration in the blood.
2. The subjects have to ingest 7 different dosages of either beetroot juice or sodium nitrate on seven different occasions. Three hours after the intake of the supplement the subjects have to perform an exercise test on a bicycle. They have to cycle 5 min at 50% of maximal oxygen consumption and 8min at 80% of maximal oxygen consumption separated by a 5min break. Oxygen consumption would be measured during the whole exercise test. Blood withdrawal is taken before the ingestion, after 3 hours and after the test.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 45
* healthy active men
* non-smoking

Exclusion Criteria:

* medication intake during study phase

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
oxygen consumption | 30min
  Oxygen consumption during exercise protocol

SECONDARY OUTCOMES:
Blood pressure | 6 hours
  every hour, blood pressure is measured.
oxygen saturation | 6 hours
  every hour oxygen saturation is measured.
Rating of perceived exertion (RPE) | during the 7 weeks of study phase
  RPE is measured after the low-intensity exercise performance and after the submaximal exercise performance.
Heart rate | during the 7 weeks of study phase
  Heart rate is measured before the ingestion, before the exercise test and during the exercise test. resting heart rate is additionally measured every hours after the intake of dietary/inorganic nitrate.
Nitrate and nitrite concentration | 6 hours
  every hour for the six hours after the ingestion of dietary/inorganic nitrate, nitrate and nitrite concentration in the blood is analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Perret, Dr. sc. nat., Principal Investigator — Sportmedizin Nottwil
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland